CLINICAL TRIAL: NCT02390713
Title: Pneumatic Reversible Portal Vein Diameter Modulation After Major Hepatectomy in Non Cirrhotic Patient
Brief Title: Pneumatic Reversible Portal Vein Diameter Modulation After Major Hepatectomy
Acronym: MODHEP1
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Medical Innovation Developpement (MID) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P131002
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Liver Failure; Major Hepatectomy
Keywords: hepatectomy; post-operative liver failure; portal vein; portal flow; portal pressure; modulation; surgical device
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MID-AVR (Experimental): Tolerance and functionality of MID-AVR during surgery (Phase A) and after surgery (Phase B)
  Interventions: Device: MID-AVR

INTERVENTIONS:
Device: MID-AVR — Phase A (4 patients): After laparotomy and dissection of hepatic pedicle, feasibility of MID-AVR positioning around the portal vein by hepato-biliary surgeon and visual evaluation of potential spatial conflict with hepatic artery and choledochal. Mid-AVR is removed at the end of surgery. Each procedure will be filmed.
  Phase B (12 patients): Mid-AVR is maintained at the end of surgery, and during 48 hours to evaluate the persistence of an hepatopetal portal flow without portal vein thrombosis upstream MID-AVR during the 48 hours after the liver surgery at bi-daily ultrasonography.

SUMMARY:
This ring aimed to preserve an intra-hepatic porto-caval gradient inferior to 5 mm Hg during and after major hepatectomy (48h) to protect the liver during the initial phases of liver regeneration. Morphological features of MID-AVRTM allow its intra corporeal opening and percutaneously removal after an balloon inflation with 5 ml of physiological serum. MID-AVRTM had been developed in pig where it had proved its efficiency to improve liver function after 75% hepatectomy and its capacity to be removed percutaneously. Aim of this feasibility study (Phase I/II) is to prove in series of 3 evaluable patients (Phase A) then 6 evaluable patients (Phase B) that MID-AVRTM could be used in human without deleterious consequence. In phase A, MID-AVRTM is dispose around the portal vein before and during a major hepatectomy performed on healthy liver and removed before abdominal closure. If phase A results confirmed that MID-AVRTM well modulates portal pressure and is easily opened and removed by acute inflation, the phase B will be started. In phase B, MID-AVRTM will be dispose around the portal vein before major hepatectomy on healthy liver and conserved 48 hours before to be removed percutaneously at the operating room.

DETAILED DESCRIPTION:
Preserving liver function is vital, especially after hepatectomy, the main curative treatment of liver tumor. An hepatectomy that preserved a remnant liver volume < 0.5% of the body weight is associated with a very high risk of post-operative liver failure. In such situation, liver volume is not sufficient to support local hemodynamic consequences of the hepatectomy that is responsible of intrahepatic endothelial cell injury that impaired liver function and regeneration. To date, preoperative vein embolization (PVE) associated or not to liver transection (ALPSS procedure) that increased future remnant liver from 20% to 90% is the only method to prevent this complication. Even this preparation is necessary for the moment, PVE increased cancer cell proliferation and is associated with lower recurrence free survival than without PVE. Despite a potential PVE, POLF occurred in 5% to 7% after major hepatectomy and stayed the first cause of death after hepatectomy. It has been demonstrated that portal pressure superior to 20 mm Hg and/or porto-caval gradient superior to 12 mm Hg at the end of hepatectomy was associated to the occurrence of POLF. Aim to avoid this acute intra hepatic portal hypertension associated to major hepatectomy that is associated with an early liver endothelial cell injury, we had developed an silicon ring to dispose around the portal vein that contained an circular inflatable balloon to narrow precisely the portal vein lumen (MID-AVRTM).

Phase A: Tolerance and functionality of MID-AVR during surgery Each procedure will be filmed. Phase B: Tolerance and functionality of MID-AVR after surgery Each procedure will be filmed.

ELIGIBILITY:
Inclusion Criteria:

* French resident affiliated to Social Insurance
* Major hepatectomy (Phase A)
* Major hepatectomy that preserved only one hepatic vein (Phase B)
* Remnant liver volume > 0.5% of the body weight

Exclusion Criteria:

* Age > 80 (Phase A) and Age > 70 (Phase B)
* Cirrhotic patient (F4)
* Repeat hepatectomy
* Patient who required a portal vein resection
* History of deep venous thrombosis
* History of portal thrombosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-04-18 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Success of MID-AVR positioning | intraoperative
  Phase A: Feasibility of MID-AVR positioning around the portal vein by hepato-biliary surgeon and visual evaluation of potential spatial conflict with hepatic artery and choledochal. Each procedure will be filmed.
Persistence of an hepatopetal portal flow at bi-daily ultrasonography | during the 48 hours after the liver surgery
  Phase B: Persistence of an hepatopetal portal flow without portal vein thrombosis upstream MID-AVR

SECONDARY OUTCOMES:
Portal pressure measured upstream and downstream the MID-AVR | intraoperative
  Phase A
Portal flow measured downstream the MID-AVR | intraoperative
  Phase A
Liver perfusion assessed by intraoperative contrast enhanced ultrasonography | intraoperative
  Phase A
Reliability of MID-AVR opening by balloon inflation and removal from the portal vein by smooth traction on the tube that is connected to MID-AVR. | intraoperative
  Phase A Each procedure will be filmed.
Occurrence of POLF (Bilirubin > 50 µmol/L and PT < 50% ) | at postoperative day 3
  Phase B
Occurrence of post-operative hemorrhage (decrease in haemoglobin that required red pack cell transfusion) | at postoperative day 3
  Phase B
Occurrence of Post-operative biliary fistulae (Bilirubin concentration in fluid drainage greater than 3 fold the plasmatic bilirubin rate) | at postoperative day 3
  Phase B
Reliability of MID-AVR opening by balloon inflation and percutaneously removal from the portal vein by smooth traction on the tube that is connected to MID-AVR. | at postoperative day 3
  Phase B Removal will be done at the operating room under neurolept analgesia and local anesthesia under radiological control. Each procedure will be filmed.

CONTACTS AND LOCATIONS:
Overall Officials: Eric VIBERT, MD, PhD, Principal Investigator — AP-HP, Paul Brousse Hospital, Centre Hepato-Biliaire, Villejuif, France
Locations (1):
- AP-HP, Paul Brousse Hospital, Centre Hepato-Biliaire, Villejuif, France